CLINICAL TRIAL: NCT02118870
Title: Randomized Evaluation of Short-term DUal Anti Platelet Therapy in Patients With Acute Coronary Syndrome Treated With the COMBO Dual-therapy stEnt
Brief Title: Short-term Dual Anti Platelet Therapy in Patients With ACS Treated With the COMBO Dual-therapy Stent
Acronym: REDUCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9207; 2013-005571-40 (EudraCT Number); 14.0102 (Other: Ethical Committee)
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS patients; Older than 18 years; PCI; Combo stent
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Therapeutics; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Aspirin; Ticagrelor; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAPT 360 days (Active Comparator): Treatment 360 days DAPT
  Interventions: Drug: Treatment 360 days DAPT
- DAPT 90 days (Active Comparator): Treatment 90 days DAPT
  Interventions: Drug: Treatment 90 days DAPT

INTERVENTIONS:
Drug: Treatment 90 days DAPT — Short term DAPT arm: will continue DAPT with P2Y12 inhibitors and ASA up to 90 days, after which patients will continue.
  Other Names: Subjects will be treated with Aspirin and P2Y12 inhibitor. Prasugrel (10; mg/day) or Ticagrelor (180 mg/day) are strongly recommended as compared; to Clopidogrel (75 mg/day)).; Short term DAPT arm: will continue DAPT with P2Y12 inhibitors and ASA up; to 90 days, after which patients will continue.
  Arms: DAPT 90 days
Drug: Treatment 360 days DAPT — Long term (360 days) DAPT arm: will continue DAPT with P2Y12 inhibitors and ASA up to 360 days, after which patients will continue on monotherapy with ASA only, unless contraindications for ASA emerge
  Other Names: Subjects will be treated with Aspirin and P2Y12 inhibitor. Prasugrel (10; mg/day) or Ticagrelor (180 mg/day) are strongly recommended as compared; to Clopidogrel (75 mg/day)).; Long term (360 days) DAPT arm: will continue DAPT with P2Y12 inhibitors and ASA up; to 360 days, after which patients will continue on monotherapy with ASA; only, unless contraindications for ASA emerge
  Arms: DAPT 360 days

SUMMARY:
Background:

The optimal duration of dual antiplatelet therapy in ACS patients treated with DES is still under debate. This is especially true for STEMI patients in the era of new anticoagulants and antiplatelet agents. Yet, the potential benefits of longterm dual antiplatelet therapy in avoiding thrombotic complications may be clearly counterbalanced by a higher risk of major bleeding complications. In particular, the COMBO dual therapy stent, being associated with early re-endothelization, may allow for a reduction of the duration of DAPT (dual anti plateled therapy) without increasing the thrombotic risk, while reducing the risk of severe bleeding complications.

Study Objective:

Aim of the current study is to demonstrate a non-inferiority of a strategy of short-term DAPT (90 days) as compared to standard 360 days DAPT in ACS patients treated with Combo stent.

Study Design:

This study is a prospective, multicenter, randomized, investigator-initiated study designed to enroll 1500 patients with ACS receiving a COMBO dual-therapy stent who will be randomized 1:1 to either short term (90 days) or to standard (360 days) DAPT. Patients will be randomized within hospitalization (before discharge in case additional revascularization is deemed necessary and performed during hospitalization). Clinical visit is scheduled at 90, and 360 days, whereas a telephone contact will be performed at 180 and 720 days.

Patient Population:

The study population will consist of up to 1500 ACS patients (male and female) older than 18 years amenable to percutaneous treatment and treated with a COMBO stent. Subjects must meet all of the eligibility criteria and provide written informed consent.

DETAILED DESCRIPTION:
Study sites:

Up to 40 investigational sites in Europe and Asia

Patients follow-up:

Follow-up (clinic) visits are scheduled at 90 and 360 days, whereas a telephone contact will be performed at 180 and 720 days. Patients randomized to short-term DAPT will continue on monotherapy with ASA after 90 days unless contraindicated.

Antiplatelet therapy:

Subjects will be treated with Aspirin and P2Y12 inhibitor. Prasugrel (10 mg/day) or Ticagrelor (180 mg/day) are strongly recommended as compared to Clopidogrel (75 mg/day)). Long term DAPT arm: will continue DAPT with P2Y12 inhibitors and ASA up to 360 days, after which patients will continue on monotherapy with ASA only, unless contraindications for ASA emerge Short term DAPT arm: will continue DAPT with P2Y12 inhibitors and ASA up to 90 days, after which patients will continue.

Timelines:

First Enrollment: June 2014 Last Enrollment: May 2016 One year Follow-up: May 2018 Two year Follow-up: May 2019

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age
2. The patient has been diagnosed with STEMI, NSTEMI or UA
3. The Patient is willing to comply with specified follow-up evaluations
4. The Patient has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics Committee (MEC), Institutional Review Board (IRB), or Human Research Ethics Committee (HREC)
5. Successful COMBO stent implantation (TIMI 3 flow with residual stenosis < 20% based visual estimation), with no clinical adverse event during hospitalization (Death, ST, stroke, TVR, bleeding (BARC II, III, V))

Exclusion Criteria:

1. Patients presenting with cardiogenic shock
2. Patients with recent major bleeding complications or contraindication to DAPT, such as:

   1. Hypersensitivity to Aspirin, Clopidogrel, Prasugrel or Ticagrelor
   2. Need for oral anticoagulation
   3. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia) or refusal of blood transfusions
   4. History of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke
   5. Stroke or transient ischemic attack within the past 6 months or any permanent residual neurologic defect
   6. Gastrointestinal or genitourinary bleeding within the last 2 months or major surgery within 6 weeks
   7. Recent history or known current platelet count <100 000 cells/mm3 or hemoglobin <10 g/dL
   8. An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 12 months post enrollment
3. Planned need for concomitant cardiac surgery (e.g., valve surgery or resection of aortic or left ventricular aneurysm etc.)
4. Planned intervention of another lesion (target vessel or non-target vessel) after index hospital discharge
5. Any revascularization performed within index hospitalization with other stents than COMBO
6. Potential for non-compliance towards the requirements in the trial protocol (especially the medical treatment) or follow-up visits
7. Patients requiring permanent DAPT due to comorbidities
8. Patient has received any organ transplant or is on a waiting list for any organ transplant
9. Life expectancy of less than 2 years
10. Pregnancy or intention to become pregnant during the course of the trial
11. Any significant medical or mental condition, which in the Investigator's opinion may interfere with the patient's optimal participation in the study
12. Currently participating in another investigational drug or device study
13. Patients who have been treated with another DES within 9 months prior to the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Composite of all cause mortality, Myocardial Infarction (MI), ST, stroke, taret vessel revascularization (TVR) and bleeding (BARC II, III and V) at 360 days | At 360 days

SECONDARY OUTCOMES:
Bleeding (BARC II, III, V) at 360 days | 360 days
All cause mortality, MI, ST, stroke, TVR, bleeding (BARC II, III, V) at 360 and 720 days | 720 days
All cause mortality, MI, ST, stroke and TVR at 360 and 720 days | 360 and 720 days
Mortality at 360 and 720 days | 360 and 720 days
Cardiac Mortality at 360 and 720 days | 360 and 720 days
Any MI at 360 and 720 days | 360 and 720 days
ST at 360 and 720 days | 360 and 720 days
Repeat revascularization at 360 and 720 days | 360 and 720 days
Time to event as defined by the occurrence of one of the following: all cause mortality, MI, ST, stroke, TVR or bleeding (BARC II, III, V) within 360 and 720 days | 360 and 720 days
Prespecified landmark analysis of Primary Endpoint (without TVR) from 90 days to 360 days | from 90 days to 360 days

CONTACTS AND LOCATIONS:
Overall Officials: H. Suryapranata, Prof. dr., Principal Investigator — Radboud University Medical Center; G. de Luca, Prof. dr., Principal Investigator — Eastern Piedmont University, Novara, Italy